CLINICAL TRIAL: NCT01186406
Title: Phase II Trial for Patients With Newly Diagnosed Glioblastoma Multiforme (GBM) Treated With Gliadel Followed by Concurrent Radiation Therapy, Temodar and Avastin, Then Followed by Avastin and Temodar Post-Radiation
Brief Title: Gliadel, XRT, Temodar, Avastin Followed by Avastin, Temodar for Newly Diagnosed Glioblastoma Multiforme (GBM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study ended early due to toxicity
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00025180
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Glioblastoma Multiforme; Gliosarcoma
Keywords: glioblastoma multiforme; gliosarcoma; malignant glioma; glioma; Gliadel; carmustine wafers; Avastin; bevacizumab; Temodar; temozolomide; Pro00025180; Desjardins; Duke; Preston Robert Tisch Brain Tumor Center
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma | interventions — carmustine, poliferprosan 20 drug combination; Carmustine; Radiotherapy; Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gliadel, Radiation Therapy, Avastin, Temodar (Experimental): Single arm study where patients with newly diagnosed Grade IV malignant glioma will receive Gliadel at the time of resection, followed by radiation therapy (XRT), Avastin, and Temodar for approximately 6 1/2 weeks, followed by Avastin and Temodar post-radiation
  Interventions: Drug: Gliadel; Radiation: Radiation Therapy; Drug: Avastin; Drug: Temodar

INTERVENTIONS:
Drug: Gliadel — Patients will have 1-8 wafers of Gliadel inserted at the time of surgical resection.
  Other Names: Gliadel (carmustine wafers)
Radiation: Radiation Therapy — At a minimum of four weeks, but not greater than eight weeks post-craniotomy, subjects will be treated with standard radiation therapy.
Drug: Avastin — Avastin (10 mg/kg) will be given every 14 days, and will begin a minimum of 42 days post-operatively.
  Beginning two to three weeks after the last radiation therapy, but not greater than eight weeks, subjects will be treated with Avastin (10mg/m2) every 14 days.
  Other Names: Avastin (bevacizumab)
Drug: Temodar — At a minimum of four weeks, but not greater than eight weeks post-craniotomy, subjects will be treated with standard radiation therapy and daily Temodar (75mg/m2) for 6.5 weeks of the radiation. In addition, beginning 2-3 weeks after the last radiation therapy, but not greater than 8 weeks, patients will be treated with 5 day Temodar (200 mg/ m2).
  Other Names: Temodar (temozolomide)

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of Gliadel wafers at the time of surgery, followed by the combination of radiation, Temodar, and Avastin, and then the combination of Avastin and Temodar, after radiation is complete, on malignant brain tumors.

About six weeks after surgery, subjects will begin standard radiation therapy, a fixed dose of Avastin every 2 weeks, and daily Temodar for the six and a half weeks of radiation. Beginning 2-3 weeks after the last radiation therapy, subjects will be given the same fixed dose of Avastin intravenously (through the vein) every 14 days. They will also be given a higher dose of oral Temodar to take daily the first 5 days of each 28-day study cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a MRI consistent with a WHO grade IV primary malignant glioma (glioblastoma multiforme or gliosarcoma), and be candidates for surgical resection with Gliadel wafer placement. Patients have to be within 6 weeks of the last major surgical procedure.
* Age ≥ 18 years
* Candidates for Gliadel
* If a prior procedure was done, an interval of at least 2 weeks and not > 8 weeks between prior major surgical procedure and study enrollment
* No prior radiotherapy or chemotherapy for a brain tumor
* Karnofsky > 60%
* Hemoglobin ≥ 9.0 g/dl, ANC ≥ 1,500 cells/microliters, platelets ≥ 125,000 cells/microliters
* Serum creatinine ≤ 1.5 mg/dl, serum SGOT and bilirubin ≤ 1.5 times upper limit of normal.
* Signed informed consent approved by the Institutional Review Board
* If sexually active, patients must agree to use appropriate contraceptive measures for the duration of the study and for 6 months afterwards as stated in the informed consent.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids.
* Active infection requiring IV antibiotics.
* Prior treatment with radiotherapy or chemotherapy for a brain tumor, irrespective of the grade of the tumor.
* Evidence of > grade 1 CNS hemorrhage on baseline MRI or CT scan.
* Prior treatment with Avastin for any condition
* Prior, unrelated malignancy requiring active treatment with the exception cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin

Avastin-Specific Exclusion Criteria:

* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study enrollment
* History of hemoptysis (≥ ½ teaspoon of bright red blood per episode) within 1 month prior to study enrollment
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first Avastin infusion or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation within 6 months prior to study enrollment
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria at screening as demonstrated by urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of Avastin
* Pregnant (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06-16 (Actual); Study Completion 2014-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Cancer Center — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment was stopped early due to unacceptable toxicity after 41 participants were enrolled.
Pre-assignment Details: Forty-seven subjects were consented to the study. Six subjects were screen failures and were not enrolled.
Groups:
- Gliadel, Radiation Therapy, Avastin, Temodar: Single arm study where patients with newly diagnosed Grade IV malignant glioma will receive Gliadel at the time of resection, followed by radiation therapy (XRT), Avastin, and Temodar for approximately 6 1/2 weeks, followed by Avastin and Temodar post-radiation
  Gliadel, Radiation Therapy, Avastin, Temodar: Patients will have 1-8 wafers of Gliadel inserted at the time of surgical resection. At a minimum of four weeks, but not greater than eight weeks post-craniotomy, they will be treated with standard radiation therapy, and daily Temodar (75mg/m2) for 6.5 weeks of radiation. In addition, Avastin (10 mg/kg) will be given every 14 days, and will begin a minimum of 42 days post-operatively.
  Beginning 2-3 weeks after the last radiation therapy, but not greater than 8 weeks, patients will be treated with Avastin (10 mg/kg) every 14 days along with 5 day Temodar (200 mg/ m2).
Period: Overall Study
Arm/Group | Gliadel, Radiation Therapy, Avastin, Temodar
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Gliadel, Radiation Therapy, Avastin, Temodar: Single arm study where patients with newly diagnosed Grade IV malignant glioma will receive Gliadel at the time of resection, followed by radiation therapy (XRT), Avastin, and Temodar for approximately 6 1/2 weeks, followed by Avastin and Temodar post-radiation Patients will have 1-8 wafers of Gliadel inserted at the time of surgical resection. At a minimum of four weeks, but not greater than eight weeks post-craniotomy, subjects will be treated with standard radiation therapy. Avastin (10 mg/kg) will be given every 14 days, and will begin a minimum of 42 days post-operatively. Beginning two to three weeks after the last radiation therapy, but not greater than eight weeks, subjects will be treated with Avastin (10mg/m2) every 14 days. At a minimum of four weeks, but not greater than eight weeks post-craniotomy, subjects will be treated with standard radiation therapy and daily Temodar (75mg/m2) for 6.5 weeks of the radiation.
Arm/Group | Gliadel, Radiation Therapy, Avastin, Temodar
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: 21-month Overall Survival
Description: The percentage of participants alive at 21 months after the start of study treatment. Overall survival was calculated from the date study treatment started until the date of death or the date of last follow-up if alive. Kaplan-Meier methods were used to estimate overall survival.
Time Frame: 21 months
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Gliadel, Radiation Therapy, Avastin, Temodar: Single arm study where patients with newly diagnosed Grade IV malignant glioma will receive Gliadel at the time of resection, followed by radiation therapy (XRT), Avastin, and Temodar for approximately 6 1/2 weeks, followed by Avastin and Temodar post-radiation. Patients will have 1-8 wafers of Gliadel inserted at the time of surgical resection. At a minimum of four weeks, but not greater than eight weeks post-craniotomy, subjects will be treated with standard radiation therapy. Avastin (10 mg/kg) will be given every 14 days, and will begin a minimum of 42 days post-operatively. Beginning two to three weeks after the last radiation therapy, but not greater than eight weeks, subjects will be treated with Avastin (10mg/m2) every 14 days. At a minimum of four weeks, but not greater than eight weeks post-craniotomy, subjects will be treated with standard radiation therapy and daily Temodar (75mg/m2) for 6.5 weeks of the radiation.
Arm/Group | Gliadel, Radiation Therapy, Avastin, Temodar
Number analyzed (Participants) | 41
percentage of participants | 40.9 [25.8 to 55.5]

2. Secondary Outcome: Median Overall Survival
Description: Overall survival was defined as the time in months from the start of SRS to the date of death or last contact if alive. Kaplan-Meier methods were used to estimate overall survival.
Time Frame: 21 months
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gliadel, Radiation Therapy, Avastin, Temodar
Number analyzed (Participants) | 41
months | 19.4 [16.1 to 21.9]

3. Secondary Outcome: Median Progression-free Survival
Description: Progression-free survival was defined as the time in months from the date study treatment started until the date of progression or the date of death if death occurred before progression, or until the date of last follow-up if alive without progression. Kaplan-Meier methods were used to estimate progression-free survival.
Time Frame: 21 months
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gliadel, Radiation Therapy, Avastin, Temodar
Number analyzed (Participants) | 41
months | 11.3 [9.2 to 14.2]

4. Secondary Outcome: Unacceptable Toxicity Related to the Treatment Regimen
Description: The number of patients experiencing unacceptable toxicity defined as the occurrence of ≥ grade 2 CNS hemorrhage or treatment-related grade 4 or 5 non-hematologic toxicity.
Time Frame: 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gliadel, Radiation Therapy, Avastin, Temodar
Number analyzed (Participants) | 41
Participants | 6.0

ADVERSE EVENTS:
Time Frame: From the start of study treatment for a patient until 30 days after treatment is discontinued.
Description: Patients will be evaluated for adverse events (all grades), serious adverse events, and adverse events requiring study drug interruption or discontinuation at each study visit for the duration of their participation. After evaluation, all adverse events graded 3 and above, and all serious adverse events will be captured in the study database.
Arm/Group | Gliadel, Radiation Therapy, Avastin, Temodar
Serious Adverse Events (participants affected / at risk) | 18/41
Other Adverse Events (participants affected / at risk) | 18/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gliadel, Radiation Therapy, Avastin, Temodar (N=41)
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 3
Edema cerebral (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 6
Stroke (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Thromboembolic event (Vascular disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gliadel, Radiation Therapy, Avastin, Temodar (N=41)
Fatigue (General disorders) | 2
Meningitis (Infections and infestations) | 1
Tooth Infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 2
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 5
White blood cell decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Psychosis (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes